CLINICAL TRIAL: NCT04800380
Title: Edpuzzle Implementation in Improving the Metric and Drug Dose Calculation Skills of Nursing Students in a Virtual Flipped Learning Environment: A Randomized Controlled Study
Brief Title: Edpuzzle Application in Improving Metric and Drug Dose Calculation Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Instructor- Principal investigator, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 440
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Nursing Students
Keywords: Nursing students; Drug; Drug dose calculation; Edpuzzle; Metric conversion account; Flipped learning

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial in parallel groups
Who Masked: Participant, Investigator
Masking Description: In the study, randomization and evaluation of results will be carried out by an independent statistician. Researchers will not know to which group the students are included. In conducting the research, an independent researcher will know in which group the students are. Students will also be given information about the study, but not in which group they are included. Thus, triple blinding will be created by providing both participant, entrepreneur and statistician blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine training (No Intervention): Nursing students in the control group will receive training in routine metric and drug dose calculation in virtual environment.
- Edpuzzle application (Experimental): Students in the intervention group will watch the routine metric and drug dose calculation training in virtual environment, as well as interactive videos prepared by the first researcher and uploaded to the Edpuzzle application.
  Interventions: Other: Edpuzzle interactive videos

INTERVENTIONS:
Other: Edpuzzle interactive videos — The effectiveness of the Edpuzzle application will be evaluated in developing the metric and drug dose calculation skills of first year nursing students.
  Arms: Edpuzzle application

SUMMARY:
This experimental, triple-blind, randomized controlled study was planned to evaluate the effect of Edpuzzle application on the metric and drug dose calculation skills of nursing students. First-year nursing students who take the Basic Principles and Practices in Nursing II course, in which metric and drug dose calculation skills are taught, will form the universe of the research. "Metric and Drug Dose Calculation Knowledge Test" will be used to evaluate students' metric and drug dose calculation skills. "Semi-Structured Focus Group Interview Form" will be used to evaluate students' views about Edpuzzle application.

DETAILED DESCRIPTION:
Study design; It is an experimental, triple blind, randomized controlled study in parallel groups.

Study population and sample: The study population in Turkey studying at a state university of Health Sciences Faculty in Central Anatolia will create first-class nursing students. The research will be carried out within the scope of this course since the metric and drug dose calculation skills are explained in the subject curriculum of Basic Principles and Applications in Nursing II. Students who meet the criteria for inclusion in the study within the universe (students enrolling in the Basic Principles and Practices in Nursing II course for the first time and willing to participate in the study voluntarily) will be randomly assigned to the control and intervention groups according to their entrance points and gender by an independent statistician. It is expected that there will be approximately 100 students who meet the criteria for inclusion in the study. 50 of these will constitute the control group and 50 of them will constitute the intervention group. Researchers will not be informed about which group the students are assigned to. In the virtual classroom environment, the first researcher will explain the metric and drug dose calculation skills within the scope of the drug applications in the course curriculum to all students, and sample questions will be solved. After the virtual classroom training, the "Metric and Drug Dose Knowledge Test" consisting of 20 closed-ended questions developed by the researchers and expert opinions will be used in the pre-test application to evaluate the metric and drug dose calculation skills of the students. Before the test is applied, students will be informed that there will be a test for metric and drug dose calculations. The test will be provided to all students who will be uploaded to the university's distance education system to enter the system at the same time and answer 20 questions in equal time. After the pre-test application, the necessary introduction information will be sent to the intervention group students to watch the interactive videos prepared by the first researcher and uploaded to the Edpuzzle application by an independent researcher. Students will be able to watch interactive videos over and over again by entering the system with their names. Questions prepared by the researchers and expert opinions were placed between interactive videos. If the student answers the question correctly, the video will continue. Thus, active participants of the videos will be provided. Edpuzzle application can provide detailed documentation of the steps each student followed in each video. After all of the students in the intervention group watch the videos, all students will be informed that they will be tested for metric and drug dosage calculations. The "Metric and Drug Dose Calculation Knowledge Test" used in the pre-test application will be loaded in the virtual exam system of the university where the study is performed again, and each student will be able to answer the questions at the same time and in equal time. Thus, the final test data will be obtained. After the pre-test and post-test applications are completed, the list of the students will be given to the researchers by the researcher, who is independent of the study and who is aware of the intervention group students, in order to get student opinions about the Edpuzzle application. With the "Semi-Structured Focus Group Interview Form" prepared by the researchers and receiving expert opinions, the students will be divided into groups of 7 and focus group interviews will be held.

ELIGIBILITY:
Inclusion Criteria:

* Enrolling in the Basic Principles and Practices in Nursing II course for the first time,
* Students who volunteer to participate in research.

Exclusion Criteria:

* Graduated from a health-related high school or university,
* Having difficulty in speaking and understanding Turkish,
* Students who do not have enough internet.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Metric and Drug Dose Calculation Knowledge Test | 2 month
  The test was prepared by the researchers to evaluate the metric and drug dose calculation knowledge of the control group students who received routine training and the intervention group students who watched Edpuzzle interactive videos. Knowledge test consists of closed-ended, five options and 20 questions. Each correct answer will count as 5 points. Thus, students will be able to get a minimum of "0" points and a maximum of "100" points from the test. It will be interpreted that as the number of questions answered correctly by the students, that is, as they approached 100 points, their level of knowledge increased.

CONTACTS AND LOCATIONS:
Overall Officials: YADİGAR ORDU, Principal Investigator — Çankırı Karatekin University; SAKINE YILMAZ, Study Chair — Çankırı Karatekin University; GÖZDE ÖZARAS ÖZ, Study Chair — Çankırı Karatekin University
Locations (1):
- Cankırı Karatekin University, Çankırı, Çankırı, Turkey (Türkiye)